CLINICAL TRIAL: NCT01295619
Title: A Prospective, Open, Multi-center, Single-arm Study of the Performance and Safety of I-020805 in the Prevention of Cerebrospinal Fluid Leakage Following Elective Cranial Surgery
Brief Title: Performance and Safety of I-020805 in Prevention of Cerebrospinal Fluid (CSF) Leakage Following Elective Craniotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CS I-020805/01
Record Dates: First submitted 2011-02-09; First posted 2011-02-14 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Cerebrospinal Fluid Leakage
Keywords: Dura; Sealant; Cranial; Craniotomy; CSF leakage; CSF leakage following cranial surgery
MeSH Terms: conditions — Cerebrospinal Fluid Leak; Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I-020805 (Experimental): This was a prospective, open, multi-center, single-arm study to investigate I-020805 in patients following elective cranial surgery. If they met the inclusion/ exclusion criteria, they receive I-020805 after suturing of the dura. If necessary, autologous grafts were to be used to augment dural closure.
  Interventions: Device: I-020805

INTERVENTIONS:
Device: I-020805 — A thin layer of I-020805 applied up to two times on the sutured dura mater

SUMMARY:
This is a prospective study to evaluate the performance and safety of a new medical device used in case of cerebrospinal fluid (CSF) leakage after an elective cranial surgery.

DETAILED DESCRIPTION:
Patients who consented to participate in the trial and fulfilled the preoperative inclusion and exclusion criteria underwent screening prior to surgical treatment. After dural suturing, if patients met the intra operative inclusion and exclusion criteria, they received I-020805. If necessary, autologous grafts were to be used to augment dural closure.

I-020805 was delivered from a double syringe applicator that creates a fine layer over the dura. This layer quickly sets within seconds to form a watertight seal.

ELIGIBILITY:
Inclusion Criteria:

Pre-operative

* Male or female of 18 years old or over
* Elective cranial procedure entailing a dural incision of at least 2 cm in length
* Requires a procedure involving surgical wound classification Class I/Clean
* Signed informed consent form
* Negative pregnancy test at screening for women of childbearing potential and agreeing to use an acceptable birth control method or abstinence until 90 days post-surgery

Intra-operative

* Surgical wound classification Class I/Clean
* Dural margin from bony edges of at least 3 mm throughout
* Spontaneous expression of CSF assessed visually or a CSF leakage upon Valsalva maneuver

Exclusion Criteria:

Pre-operative

* Cranial procedure requiring translabyrinthine, transoral and/or any procedure penetrating the air sinus or mastoid air cells
* Presence of symptomatic hydrocephalus
* Pre-existing external ventricular drainage or lumbar CSF drain
* Radiotherapy in the planned surgical region which ended within 3 months prior to planned surgery
* Presence of systemic infection
* Known history of hemophilia or other clinically significant coagulopathy
* Known oral anticoagulant use
* Pregnancy or breast feeding
* Known allergy to any components of I-020805
* Previous participation in this trial or any investigational drug or device study within 30 day of screening
* Known clinically significant organ or systemic diseases
* Known or suspected non-compliance with trial procedures

Intra-operative

* Patient not meeting the pre-operative eligibility criteria
* Not able to tolerate a Valsalva maneuver
* Gap of more than 2 mm remaining after primary closure of dura
* Use of synthetic or non-autologous duraplasty material

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Performance of I-020805 in prevention of CSF leakage | Intraoperative on the day of sugery

SECONDARY OUTCOMES:
Incidence of CSF leakage | Within 7 days after surgery or prior to discharge
CSF leakage or pseudomeningocele related surgical intervention | Within 90 days following surgery
CSF leakage confirmed by clinical evaluation or diagnostic testing | Within 90 days following surgery
Surgical infection and unexpected neurological signs | Post-operative and within 7 days and 90 following surgery
Wound healing impairment | Throughout study up to 90 days following surgery
Incidence of all and treatment emergent adverse events | Throughout study up to 90 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Jamieson, MD, Study Director — Kuros Biosurgery
Locations (4):
- Charite Universitätsmedizin (01), Berlin, Germany
- Hungary (3):
  - Orszagos Idegtudomanyi Intezet (11), Budapest
  - Debreceni Tudomanyegyetem (12), Debrecen
  - Szegedi Tudomanyegyetem (10), Szeged

IPD SHARING:
Plan to Share IPD: No